CLINICAL TRIAL: NCT07057934
Title: THE EFFECTS OF EXTERNAL OBLIQUE INTERCOSTAL PLAN BLOCK AND ERECTOR SPINA PLAN BLOCK ON POSTOPERATIVE ANALGESIA IN PATIENTS UNDERGOING LAPAROSCOPIC CHOLECYSTECTOMY OPERATION
Brief Title: Comparative Efficacy of ESPB and EOPB for Postoperative Analgesia in Laparoscopic Cholecystectomy: A Randomized Controlled Trial (External Oblique Intercostal Plan Block (EOPB) and Erector Spina Plan Block (ESPB) )
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Dr. Lutfi Kirdar Kartal Training and Research Hospital (Other Government)
Responsible Party: Principal Investigator, Aykut Aydin, M.D., Dr. Lutfi Kirdar Kartal Training and Research Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: SBÜ-KLKH-AR-2024-ESPB-EOPB-01; 2024/17/840-938 (Other: Ethics Committee Reference Number)
Record Dates: First submitted 2025-06-30; First posted 2025-07-10 (Actual); Last update posted 2025-07-10 (Actual); Status verified 2025-06

CONDITIONS: Postoperative Pain; Cholelithiasis; Acute Pain
Keywords: Laparoscopic Cholecystectomy; Regional Anesthesia; Erector Spinae Plane Block; External Oblique Intercostal Plane Block; Multimodal Analgesia
MeSH Terms: conditions — Pain, Postoperative; Cholelithiasis; Acute Pain

STUDY DESIGN:
Intervention Model Description: This is a single-center, prospective, randomized, controlled, parallel-group clinical trial involving 90 patients undergoing elective laparoscopic cholecystectomy under general anesthesia. Participants were randomly allocated into three groups:
  ESPB Group: Patients received a bilateral erector spinae plane block at the T7-T8 level prior to surgical incision.
  EOPB Group: Patients received an external oblique intercostal plane block at the 6th rib level.
  Control Group: Patients received no regional block. All participants were monitored for postoperative pain scores and analgesic consumption over 24 hours.
Who Masked: Participant, Care Provider, Investigator
Masking Description: The local anesthetic to be used in the study was prepared by two researchers who were not involved in the anesthesia application and did not participate in the postoperative data collection process. Postoperative patient data were recorded with the random ID assigned to each patient, and the researchers who collected data during this process were not informed about the patient groups. In addition, the anesthesiologist who performed the simple randomization also performed the nerve block, but was not involved in the collection of postoperative data. The anesthesiologists responsible for the anesthesia management and data collection process were not informed about the group distribution, and thus the study was conducted in a double-blind manner.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Erector Spinae Plane Block (ESPB) (Experimental): Participants in this group received a bilateral ultrasound-guided erector spinae plane block (ESPB) at the T7-T8 vertebral level under general anesthesia prior to surgical incision.
  Under sterile conditions and ultrasound guidance, 20 mL of local anesthetic solution (10 mL of 0.5% bupivacaine and 10 mL of 2% lidocaine) was injected bilaterally into the erector spinae plane at the T7-T8 level before incision. The block was performed after induction of general anesthesia but before the start of laparoscopic cholecystectomy.
  Interventions: Procedure: ESPB Block
- External Oblique Intercostal Plane Block (EOPB) (Experimental): Participants in this group received an external oblique intercostal plane block (EOPB) under ultrasound guidance prior to surgical incision.
  Under ultrasound guidance, 20 mL of local anesthetic mixture (10 mL of 0.5% bupivacaine and 10 mL of 2% lidocaine) was injected into the fascial plane between the external oblique and internal intercostal muscles at the level of the 6th rib. The procedure was done after anesthesia induction but prior to laparoscopic cholecystectomy.
  Interventions: Procedure: EOPB Block
- Control Group (Other): Participants in this group did not receive any regional block. Postoperative analgesia was provided via standard systemic medications as needed.
  No regional anesthesia technique was applied. Postoperative pain was managed using systemic rescue analgesia: 50 mg dexketoprofen trometamol IV when VAS ≥4, followed by 50 mg tramadol IV if pain persisted.
  Interventions: Drug: Standard Systemic Analgesia

INTERVENTIONS:
Procedure: ESPB Block — Under sterile conditions and ultrasound guidance, 20 mL of local anesthetic solution (10 mL of 0.5% bupivacaine and 10 mL of 2% lidocaine) was injected bilaterally into the erector spinae plane at the T7-T8 level before incision. The block was performed after induction of general anesthesia but before the start of laparoscopic cholecystectomy.
  Arms: Erector Spinae Plane Block (ESPB)
Procedure: EOPB Block — Under ultrasound guidance, 20 mL of local anesthetic mixture (10 mL of 0.5% bupivacaine and 10 mL of 2% lidocaine) was injected into the fascial plane between the external oblique and internal intercostal muscles at the level of the 6th rib. The procedure was done after anesthesia induction but prior to laparoscopic cholecystectomy.
  Arms: External Oblique Intercostal Plane Block (EOPB)
Drug: Standard Systemic Analgesia — No regional anesthesia technique was applied. Postoperative pain was managed using systemic rescue analgesia: 50 mg dexketoprofen trometamol IV when VAS ≥4, followed by 50 mg tramadol IV if pain persisted.
  Arms: Control Group

SUMMARY:
This randomized controlled clinical trial investigates the comparative efficacy of two novel regional anesthesia techniques - the Erector Spinae Plane Block (ESPB) and the External Oblique Intercostal Plane Block (EOPB) - for postoperative analgesia in patients undergoing elective laparoscopic cholecystectomy under general anesthesia.

A total of 90 patients aged 18-65 years, with ASA physical status I or II, were randomly assigned to one of three groups: ESPB, EOPB, or control. Blocks were performed under ultrasound guidance prior to surgical incision. Pain intensity was evaluated using the Visual Analog Scale (VAS), and rescue analgesic consumption was recorded over the first 24 hours postoperatively.

The study aims to determine whether ESPB or EOPB offers superior pain control and reduced opioid consumption, and to assess patient satisfaction and safety. The results will inform multimodal analgesia strategies for upper abdominal laparoscopic surgery.

DETAILED DESCRIPTION:
Laparoscopic cholecystectomy (LC) is one of the most commonly performed upper abdominal surgeries. Despite being minimally invasive, LC is frequently associated with significant postoperative pain originating from both visceral and somatic sources. Inadequate pain control may lead to delayed recovery, increased opioid consumption, and patient dissatisfaction.

Regional anesthesia techniques have become increasingly important components of multimodal analgesia protocols for abdominal surgeries. Two recently described fascial plane blocks - the Erector Spinae Plane Block (ESPB) and the External Oblique Intercostal Plane Block (EOPB) - have shown promising results in reducing postoperative pain in thoracic and abdominal procedures.

This prospective, randomized, controlled clinical trial was conducted to evaluate and compare the analgesic effectiveness of ESPB and EOPB in patients undergoing elective LC under general anesthesia. After obtaining ethical approval (Protocol No: 2024/17/840-938) and informed consent, 90 adult patients aged 18-65 years with ASA physical status I or II were enrolled.

Participants were randomized into three groups using a sealed envelope technique:

Group 1 (ESPB): Received bilateral ultrasound-guided ESPB at the T7-8 level using 20 mL of local anesthetic solution (10 mL 0.5% bupivacaine + 10 mL 2% lidocaine) preoperatively.

Group 2 (EOPB): Received ultrasound-guided EOPB using the same volume and mixture of local anesthetic.

Group 3 (Control): Did not receive any regional block.

Postoperative pain was assessed using the Visual Analog Scale (VAS) at regular intervals (15 minutes, and at 2, 4, 8, 12, 16, and 24 hours). Rescue analgesia consisted of 50 mg dexketoprofen trometamol administered when VAS ≥4. If pain persisted, 50 mg tramadol was given as a second-line analgesic.

Primary endpoints included postoperative VAS scores and total rescue analgesic consumption over 24 hours. Secondary endpoints included time to first analgesic requirement, side effects, complications related to blocks, and patient satisfaction.

Initial results indicated that both ESPB and EOPB significantly reduced postoperative pain and analgesic requirements compared to the control group. While EOPB was technically easier to perform, ESPB provided longer-lasting analgesia. These findings may support the integration of ESPB or EOPB into routine multimodal analgesia protocols for laparoscopic abdominal surgeries.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-65 years
* ASA physical status I-II
* Undergoing elective laparoscopic cholecystectomy under general anesthesia
* Provided informed written consent
* BMI between 18.5 and 30 kg/m²
* Able to follow study instructions

Exclusion Criteria:

* Allergy to local anesthetics
* Chronic opioid use or chronic pain
* Coagulopathy or anticoagulant use
* Severe organ dysfunction
* Pregnancy or breastfeeding
* Neurological or psychiatric disorders
* Infection at injection site
* Refusal to participate

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2024-04-01 (Actual); Primary Completion 2024-06-30 (Actual); Study Completion 2024-06-30 (Actual)

PRIMARY OUTCOMES:
Postoperative Pain Intensity (VAS Score) | 0-24 hours postoperatively (measured at 15 min, 2, 4, 8, 12, 16, and 24 hours)
  Postoperative pain will be measured using the Visual Analog Scale (VAS), where patients rate their pain on a 0-10 scale (0 = no pain, 10 = worst imaginable pain).
Total Rescue Analgesic Consumption (Dexketoprofen + Tramadol) | 0-24 hours postoperatively
  Total cumulative dose of rescue analgesics administered within the first 24 hours postoperatively will be recorded. Dexketoprofen (mg) and tramadol (mg) will be summed for each participant.

SECONDARY OUTCOMES:
Time to First Rescue Analgesic Requirement | 0-24 hours postoperatively
  The time elapsed from the end of surgery to the administration of the first dose of rescue analgesic (dexketoprofen) will be recorded for each participant.
Patient Satisfaction Score | At 24 hours postoperatively
  Patient satisfaction with pain management will be assessed at 24 hours using a 5-point Likert scale (1 = very dissatisfied, 5 = very satisfied).
Incidence of Block-Related Complications | Intraoperative and within 24 hours postoperative
  Incidence of complications related to regional blocks (e.g., local anesthetic toxicity, hematoma, nerve injury, pneumothorax) will be monitored and recorded.
Intraoperative Opioid Requirement | Intraoperative period (during surgery)
  Total intraoperative fentanyl dose (in mcg) administered during the procedure will be recorded.

CONTACTS AND LOCATIONS:
Locations (1):
- Aykutaydiniu@Gmail.Com, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
Individual participant data (IPD) will not be shared. The study was conducted as part of a postgraduate academic thesis, and ethical approval limits data use to the original analysis only. No public data repository or external sharing is planned.